CLINICAL TRIAL: NCT03831997
Title: The Effect of Dextrose 5% in 0.225% Sodium Chloride (D5 1/4NS) on Postoperative Chronic Subdural Hematoma Size and Recurrence Rate
Brief Title: Effect of Different Intravenous Fluids on Post-operative Chronic Subdural Hematoma Size and Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Eric A. Marvin, Principle Investigator, Carilion Clinic
Other Study IDs: #2589
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Glucose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Historical Controls: The retrospective arm will consist of our control group, it will be derived from a retrospective medical chart review of all patients with CSDH at the facility.
- Prospective Arm: The prospective arm of the study will be looking at the effects of Dextrose 5% W/ Sodium Chloride 0.225% on the recurrence rate defined by the need for secondary surgical intervention for residual/recurrent CSDH) of CSDH in a 3-month post-operative window.
  Interventions: Drug: Dextrose 5% W/ Sodium Chloride 0.225%

INTERVENTIONS:
Drug: Dextrose 5% W/ Sodium Chloride 0.225% — D5 1/4NS is comprised of 5% dextrose in a 0.225% sodium chloride (NaCl) solution. D5 1/4NS is initially slightly hypertonic to plasma, with an osmolarity of 321 mOSm/L. As the glucose component is rapidly metabolized, 0.225% NaCl solution remains and is hypotonic to plasma at an osmolarity of 77 mOsm/L. Because of the hypotonicity of the 1/4NS, it shifts into the intracellular compartments, followed by free water, and allows for volume expansion.
  Other Names: D5 1/4NS
  Groups: Prospective Arm

SUMMARY:
This study aims to reduce the recurrence rate of chronic subdural hematomas (CSDH) by manipulating the post-operative intravenous fluid use. The hypothesis relies on the relationship between osmolality and volume changes related to osmolality. We will be administering dextrose 5% in 1/4 normal saline (D5 1/4NS) post-operatively to induce brain expansion which can take up the residual CSDH space, to help reduce recurrence rate.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is a neurological disease characterized by a collection of fluid, blood, and blood degradation matter between the arachnoid and dura mater in a well-developed membrane cavity. The presentation of this disease begins with minor head trauma and takes 4-7 weeks to become symptomatic.

One of the significant problems exists with CSDH is the rate of recurrence, which currently stands at a 7-30% rate worldwide. The recurrence of a CSDH is typically defined as the presence of residual or recurrent CSDH after the first resolution, leading to additional surgical intervention either within 3 months (early recurrence) or after 3 months (late recurrence). Additional surgical intervention (recurrence rate) is the outcome variable that our study will be looking at. Factors leading to persistent recurrence include age, use of anticoagulant therapy, volume of hematoma cavity, degree of midline shift on CT, presence of residual air post-operatively, and volume of residual hematoma fluid. The variability in surgeons' operative and post-operative care, which tries to address the multiple factors that lead to recurrence, illustrates the difficulty in trying to reduce postoperative recurrence. In fact, there is no postoperative standard of care. These variations in operative and postoperative care have yet to significantly decrease the recurrent rate of CSDH.

Given the health status and fragility of the patient population that is most commonly affected by CSDHs, and the inherent morbidity related to operating on this population, we hypothesize that D5 1/4NS can help mitigate the issue of residual/recurrence CSDH leading to subsequent surgeries. The fluid dynamics of D5 1/4NS have been studied and we can assume that it will facilitate brain re-expansion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic subdural hematoma (based on imaging)
* Need for surgical intervention (assessed by attending neurosurgeon based on full neurological assessment)
* The procedure of choice is burr hole drainage
* Cessation of anti-coagulant therapy with accompanying normal lab values in appropriate time frames respective to the drug
* Tolerance of supine position

Exclusion Criteria:

* <60 years old
* Presence of acute hemorrhage, stroke, or parenchymal damage
* Neurological deficits not accountable to mass effect
* Hyponatremia or inherent electrolyte imbalances
* Pregnancy or non-consentable patients
* Previous neurological surgery up to 1 year before being considered for the study
* Rapid re-expansion of brain observed intraoperatively by attending neurosurgeon
* Congestive heart failure or other medical conditions precluding normal postoperative administration of IV fluids
* Blood glucose levels > 135 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be recruiting patients (male, female; 18-60 years old) from our center, Carilion Roanoke Memorial Hospital, that have been diagnosed with CSDH necessitating burr-hole evacuation who fit our inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | Within 120 days (+/- 7 days) of their initial burr-hole surgery.
  We will see how many patients who are treated with D5 1/4NS have a recurrent episode of CSDH after their post-operative treatment.

SECONDARY OUTCOMES:
Rate of Volume Change of Residual CSDH Space | 24 (+/- 6 hours) hours post-operative.
  We will see how fast the brain volume expands after the administration of both NS and D5 1/4NS.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Marvin, DO, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvis-Miranda HR, Castellar-Leones SM, Moscote-Salazar LR. Intravenous Fluid Therapy in Traumatic Brain Injury and Decompressive Craniectomy. Bull Emerg Trauma. 2014 Jan;2(1):3-14. PMID 27162857
- [Background] Balser D, Farooq S, Mehmood T, Reyes M, Samadani U. Actual and projected incidence rates for chronic subdural hematomas in United States Veterans Administration and civilian populations. J Neurosurg. 2015 Nov;123(5):1209-15. doi: 10.3171/2014.9.JNS141550. Epub 2015 Mar 20. PMID 25794342
- [Background] De Bonis P, Trevisi G, de Waure C, Sferrazza A, Volpe M, Pompucci A, Anile C, Mangiola A. Antiplatelet/anticoagulant agents and chronic subdural hematoma in the elderly. PLoS One. 2013 Jul 12;8(7):e68732. doi: 10.1371/journal.pone.0068732. Print 2013. PMID 23874740
- [Background] Dickerson RN, Maish GO 3rd, Weinberg JA, Croce MA, Minard G, Brown RO. Safety and efficacy of intravenous hypotonic 0.225% sodium chloride infusion for the treatment of hypernatremia in critically ill patients. Nutr Clin Pract. 2013 Jun;28(3):400-8. doi: 10.1177/0884533613483840. Epub 2013 Apr 22. PMID 23609478
- [Background] Edlmann E, Giorgi-Coll S, Whitfield PC, Carpenter KLH, Hutchinson PJ. Pathophysiology of chronic subdural haematoma: inflammation, angiogenesis and implications for pharmacotherapy. J Neuroinflammation. 2017 May 30;14(1):108. doi: 10.1186/s12974-017-0881-y. PMID 28558815
- [Background] Fedorov A, Beichel R, Kalpathy-Cramer J, Finet J, Fillion-Robin JC, Pujol S, Bauer C, Jennings D, Fennessy F, Sonka M, Buatti J, Aylward S, Miller JV, Pieper S, Kikinis R. 3D Slicer as an image computing platform for the Quantitative Imaging Network. Magn Reson Imaging. 2012 Nov;30(9):1323-41. doi: 10.1016/j.mri.2012.05.001. Epub 2012 Jul 6. PMID 22770690
- [Background] Feldman Z, Kanter MJ, Robertson CS, Contant CF, Hayes C, Sheinberg MA, Villareal CA, Narayan RK, Grossman RG. Effect of head elevation on intracranial pressure, cerebral perfusion pressure, and cerebral blood flow in head-injured patients. J Neurosurg. 1992 Feb;76(2):207-11. doi: 10.3171/jns.1992.76.2.0207. PMID 1730949
- [Background] Janowski M, Kunert P. Intravenous fluid administration may improve post-operative course of patients with chronic subdural hematoma: a retrospective study. PLoS One. 2012;7(4):e35634. doi: 10.1371/journal.pone.0035634. Epub 2012 Apr 20. PMID 22532865
- [Background] Kirk T, Jones K, Miller S, Corbett J. Measurement of intraocular and intracranial pressure: is there a relationship? Ann Neurol. 2011 Aug;70(2):323-6. doi: 10.1002/ana.22414. Epub 2011 Jun 27. PMID 21710618
- [Background] Komotar RJ, Starke RM, Connolly ES. The role of drain placement following chronic subdural hematoma evacuation. Neurosurgery. 2010 Feb;66(2):N15-6. doi: 10.1227/01.neu.0000367840.82764.3a. No abstract available. PMID 20087120
- [Background] Matsumoto H, Hanayama H, Okada T, Sakurai Y, Minami H, Masuda A, Tominaga S, Miyaji K, Yamaura I, Yoshida Y. Which surgical procedure is effective for refractory chronic subdural hematoma? Analysis of our surgical procedures and literature review. J Clin Neurosci. 2018 Mar;49:40-47. doi: 10.1016/j.jocn.2017.11.009. Epub 2017 Dec 20. PMID 29274740
- [Background] Montano N, Stifano V, Skrap B, Mazzucchi E. Management of residual subdural hematoma after burr-hole evacuation. The role of fluid therapy and review of the literature. J Clin Neurosci. 2017 Dec;46:26-29. doi: 10.1016/j.jocn.2017.08.041. Epub 2017 Sep 5. PMID 28887078
- [Background] Motiei-Langroudi R, Stippler M, Shi S, Adeeb N, Gupta R, Griessenauer CJ, Papavassiliou E, Kasper EM, Arle J, Alterman RL, Ogilvy CS, Thomas AJ. Factors predicting reoperation of chronic subdural hematoma following primary surgical evacuation. J Neurosurg. 2018 Nov 1;129(5):1143-1150. doi: 10.3171/2017.6.JNS17130. Epub 2017 Dec 15. PMID 29243977
- [Background] Oh HJ, Lee KS, Shim JJ, Yoon SM, Yun IG, Bae HG. Postoperative course and recurrence of chronic subdural hematoma. J Korean Neurosurg Soc. 2010 Dec;48(6):518-23. doi: 10.3340/jkns.2010.48.6.518. Epub 2010 Dec 31. PMID 21430978
- [Background] Prud'homme M, Mathieu F, Marcotte N, Cottin S. A Pilot Placebo Controlled Randomized Trial of Dexamethasone for Chronic Subdural Hematoma. Can J Neurol Sci. 2016 Mar;43(2):284-90. doi: 10.1017/cjn.2015.393. Epub 2016 Feb 8. PMID 26853325
- [Background] Rohde V, Graf G, Hassler W. Complications of burr-hole craniostomy and closed-system drainage for chronic subdural hematomas: a retrospective analysis of 376 patients. Neurosurg Rev. 2002 Mar;25(1-2):89-94. doi: 10.1007/s101430100182. PMID 11954771
- [Background] Thotakura AK, Marabathina NR. Nonsurgical Treatment of Chronic Subdural Hematoma with Steroids. World Neurosurg. 2015 Dec;84(6):1968-72. doi: 10.1016/j.wneu.2015.08.044. Epub 2015 Sep 2. PMID 26342776
- [Background] Yadav YR, Parihar V, Namdev H, Bajaj J. Chronic subdural hematoma. Asian J Neurosurg. 2016 Oct-Dec;11(4):330-342. doi: 10.4103/1793-5482.145102. PMID 27695533
- [Background] Zhang Y, Chen S, Xiao Y, Tang W. Effects of Dexamethasone in the Treatment of Recurrent Chronic Subdural Hematoma. World Neurosurg. 2017 Sep;105:115-121. doi: 10.1016/j.wneu.2017.05.135. Epub 2017 May 31. PMID 28578110
- [Background] Zornow MH, Prough DS. Fluid management in patients with traumatic brain injury. New Horiz. 1995 Aug;3(3):488-98. PMID 7496759